CLINICAL TRIAL: NCT03611556
Title: A Phase 1b/2 Study to Evaluate the Safety, Pharmacokinetics, and Clinical Activity of Oleclumab (MEDI9447) With or Without Durvalumab in Combination With Chemotherapy in Subjects With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: MEDI9447(Oleclumab) Pancreatic Chemotherapy Combination Study.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6070C00005; D6070C00005 (Other Grant/Funding Number: MedImmune, LLC); 2018-001028-21 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-08-02 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Carcinoma; Metastatic Pancreatic Adenocarcinoma
Keywords: MEDI9447; oleclumab; immunotherapy; pancreatic cancer; durvalumab
MeSH Terms: conditions — Carcinoma; Pancreatic Neoplasms | interventions — durvalumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + nab-paclitaxel (Experimental): Participants with 1L metastatic disease will receive intravenous (IV) infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then every 4 weeks (Q4W) in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Durvalumab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel (Experimental): Participants with 1L metastatic disease will receive IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Durvalumab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX (Experimental): Participants with 2L metastatic disease will receive IV infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of mFOLFOX (oxaliplatin 85 mg/m^2 IV; folinic acid 400 mg/m^2 IV; 5-FU 400 mg/m^2 IV bolus followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours) on Days 1 and 15 and then repeated on a Q4W schedule, until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Durvalumab; Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-FU
- Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX (Experimental): Participants with 2L metastatic disease will receive IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of mFOLFOX (oxaliplatin 85 mg/m^2 IV; folinic acid 400 mg/m^2 IV; 5-FU 400 mg/m^2 IV bolus followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours) on Days 1 and 15 and then repeated on a Q4W schedule, until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Durvalumab; Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-FU
- Dose-expansion, Gemcitabine + nab-paclitaxel (Active Comparator): Participants with 1L metastatic disease will receive IV infusions of chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel
- Dose-expansion, Oleclumab 3000 mg + Gemcitabine + nab-paclitaxel (Experimental): Participants with 1L metastatic disease will receive IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel (Experimental): Participants with 1L metastatic disease will receive IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion is met.
  Interventions: Drug: Oleclumab; Drug: Durvalumab; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Oleclumab — Participants will receive IV infusion of oleclumab as stated in arm description.
  Other Names: MEDI9447
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX; Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX; Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Gemcitabine + nab-paclitaxel
Drug: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arm description.
  Other Names: MEDI4736
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX; Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX; Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel
Drug: Gemcitabine — Participants will receive IV infusion of gemcitabine as stated in arm description.
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-expansion, Gemcitabine + nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Gemcitabine + nab-paclitaxel
Drug: Nab-paclitaxel — Participants will receive IV infusion of nab-paclitaxel as stated in arm description.
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-expansion, Gemcitabine + nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Gemcitabine + nab-paclitaxel
Drug: Oxaliplatin — Participants will receive IV infusion of oxaliplatin as stated in arm description.
  Other Names: Modified FOLFOX (oxaliplatin, folinic acid, and 5-FU)
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX; Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Drug: Folinic acid — Participants will receive IV infusion of folinic acid as stated in arm description.
  Other Names: Modified FOLFOX (oxaliplatin, folinic acid, and 5-FU)
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX; Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Drug: 5-FU — Participants will receive IV infusion of 5-FU as stated in arm description.
  Other Names: Modified FOLFOX (oxaliplatin, folinic acid, and 5-FU)
  Arms: Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX; Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and antitumor activity of oleclumab (MEDI9447) in combination with or without durvalumab plus chemotherapy in participants with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a Phase 1b/2, multicenter, open-label, dose-escalation, and dose-expansion study to assess the safety, preliminary antitumor activity, immunogenicity, and pharmacokinetics (PK) of oleclumab with or without durvalumab in combination with chemotherapy administered in participants with metastatic pancreatic ductal adenocarcinoma (PDAC). Participants with previously untreated metastatic PDAC (first-line [1L] metastatic PDAC) will be enrolled in Cohort A. Participants with metastatic PDAC previously treated with gemcitabine-based chemotherapy (without exposure to 5-fluorouracil [5-FU], capecitabine, or oxaliplatin; second-line [2L] metastatic PDAC) will be enrolled in Cohort B. The study consists of 2 parts, dose escalation (Part 1) and dose expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18
2. Written and signed informed consent must be obtained
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
4. Weight >= 35 kg
5. Participants must have histologically or cytologically, confirmed pancreatic adenocarcinoma:

   Cohort A: Participants with previously untreated metastatic pancreatic adenocarcinoma (1L metastatic disease) not previously treated with systemic therapies Cohort B: Participants with metastatic pancreatic adenocarcinoma previously treated with gemcitabine-based chemotherapy (without exposure to 5-FU, capecitabine, oxaliplatin) 2L metastatic disease
6. Participants must have at least 1 measurable lesion according to RECIST v1.1
7. All Participants must consent to providing archival tumor specimens.

Exclusion Criteria:

1. Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 14 days prior to the scheduled first dose of study treatment.
2. Prior receipt of any immune-related therapy
3. Concurrent enrollment in another therapeutic clinical study. Enrollment in observational studies will be allowed.
4. Participants with a history of venous thrombosis within the past 3 months
5. Participants with prior history of myocardial infarction, transient ischemic attack, or stroke in the last 3 months prior to start of treatment
6. Active or prior documented autoimmune or inflammatory disorders within the past 3 years prior to the start of treatment
7. Other invasive malignancy within 2 years
8. Any history of leptomeningeal disease or cord compression
9. Current or prior use of immunosuppressive medication within 14 days prior to the first dose.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (17):
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Buffalo, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Australia (4):
  - Research Site, Blacktown
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, St Leonards
- Research Site, Oslo, Norway
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Fuenlabrada
  - Research Site, Oviedo
  - Research Site, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00005&attachmentIdentifier=0fb0e4a6-ef94-4658-9a6d-b9d2f77f571f&fileName=d6070c00005-csp-amendment-3-Redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00005&attachmentIdentifier=636c01ef-f3da-4eec-b9de-de1fe3ac4864&fileName=d6070c00005-sap-ed-3-Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00005&attachmentIdentifier=1f662c2d-1eb8-4c56-9b23-87d6bb71975d&fileName=d6070c00005-study-synopsis-Redacted-PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 25 participants were treated in dose escalation part of this study. A total of 188 participants were randomised in dose expansion part of this study of which 170 participants were treated (18 participants were randomised but not treated). Results are presented for 195 treated participants only.
Groups:
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: Participants with first-line (1L) metastatic disease received intravenous (IV) infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then every 4 weeks (Q4W) in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel; Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: Participants with 1L metastatic disease received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX: Participants with second-line (2L) metastatic disease received IV infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of mFOLFOX (oxaliplatin 85 mg/m^2 IV; folinic acid 400 mg/m^2 IV; fluorouracil [5-FU] 400 mg/m^2 IV bolus followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours) on Days 1 and 15 and then repeated on a Q4W schedule, until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX: Participants with 2L metastatic disease received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of mFOLFOX (oxaliplatin 85 mg/m^2 IV; folinic acid 400 mg/m^2 IV; 5-FU 400 mg/m^2 IV bolus followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours) on Days 1 and 15 and then repeated on a Q4W schedule, until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Dose-expansion, Gemcitabine + Nab-paclitaxel: Participants with 1L metastatic disease received IV infusions of chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: Participants with 1L metastatic disease received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Started | 7 | 7 | 3 | 8 | 62 | 38 | 70
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 3 | 8 | 62 | 38 | 70
Not completed — Death | 7 | 7 | 3 | 8 | 47 | 32 | 53
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2 | 4
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 9 | 4 | 12
Not completed — Reasons | 0 | 0 | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drugs and were analyzed according to the treatment they actually received.
Groups:
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: Participants with 1L metastatic disease received IV infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Total
Number analyzed (Participants) | 7 | 7 | 3 | 8 | 62 | 38 | 70 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (12.8) | 59.6 (11.4) | 67.0 (14.9) | 64.8 (4.8) | 65.6 (8.0) | 62.5 (11.1) | 62.9 (8.3) | 63.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 4 | 26 | 17 | 34 | 89
  Male | 4 | 3 | 2 | 4 | 36 | 21 | 36 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 7 | 7 | 3 | 7 | 61 | 37 | 69 | 191
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 2 | 3 | 2 | 2 | 10
  White | 6 | 5 | 3 | 6 | 54 | 33 | 64 | 171
  More than one race | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) in Dose Escalation Phase
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 65.7 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX: Participants with 2L metastatic disease received IV infusions of oleclumab 1500 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of mFOLFOX (oxaliplatin 85 mg/m^2 IV; folinic acid 400 mg/m^2 IV; fluorouracil [5-FU] 400 mg/m^2 IV bolus followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours) on Days 1 and 15 and then repeated on a Q4W schedule, until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Participants
  Any TEAEs | 7 | 7 | 3 | 8
  Any TESAEs | 4 | 6 | 0 | 4

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) in Dose Escalation Phase
Description: DLT: Any study drug related Grade (G)3 or higher toxicity including: any G4 immune-mediated AEs, >=G3 colitis/pneumonitis/interstitial lung disease (ILD), >=G3 nausea/vomiting/diarrhea that does not resolve to G2 or less within 3 days of maximal supportive care (MSC), G2 pneumonitis/ILD that does not resolve within 7 days of initiation of MSC, G4 anemia, G3 anemia with clinical sequelae/requires >2 units of red blood cells transfusion, G4 thrombocytopenia/neutropenia >=7 days, G3/4 thrombocytopenia with >=G3 hemorrhage, G4 febrile neutropenia (FN), G3 FN lasting >=5 days while receiving MSC, isolated G3 liver transaminase elevation (LTE)/ isolated G3 total bilirubin (TBL) that does not downgrade to G1 or less within 14 days of onset, isolated G4 LTE or TBL, elevated aspartate aminotransferase/alanine aminotransferase >3×upper limit of normal (ULN) and concurrent TBL >2×ULN without cholestasis or alternative explanations, any other toxicity judged as a DLT by Dose Escalation Committee.
Time Frame: From Day 1 to 28 days after the first dose of study drugs
Population: The DLT-evaluable population included all participants enrolled in the dose-escalation phase who received all planned doses of study drugs during the DLT evaluation period and completed the safety follow-up through the DLT evaluation period or experienced any DLT during the DLT-evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 5 | 6 | 3 | 8
Participants | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Dose Escalation Phase
Description: Number of participants with abnormal vital signs (temperature, blood pressure, pulse rate, and respiratory rate) reported as TEAEs are reported.
Time Frame: Day 1 through 65.7 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Participants
  Pyrexia | 3 | 3 | 0 | 1
  Dyspnoea | 1 | 0 | 0 | 0
  Dyspnoea exertional | 0 | 1 | 0 | 0
  Hypotension | 2 | 1 | 0 | 1
  Temperature intolerance | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs in Dose Escalation Phase
Description: Number of participants with abnormal ECG parameters reported as TEAEs are reported.
Time Frame: Day 1 through 65.7 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Participants
  Atrial fibrillation | 0 | 1 | 0 | 0
  Tachycardia | 0 | 1 | 0 | 0
  Atrioventricular block | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Dose Escalation Phase
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Time Frame: Day 1 through 65.7 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Participants
  Anaemia | 3 | 3 | 1 | 0
  Neutropenia | 2 | 2 | 2 | 1
  Thrombocytopenia | 2 | 2 | 2 | 1
  Hypothyroidism | 0 | 1 | 0 | 1
  Alanine aminotransferase increased | 3 | 4 | 0 | 2
  Aspartate aminotransferase increased | 3 | 3 | 0 | 3
  Blood alkaline phosphatase increased | 2 | 1 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0 | 1
  Blood creatinine increased | 0 | 3 | 0 | 0
  Blood glucose decreased | 1 | 0 | 0 | 0
  International normalised ratio increased | 1 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 1 | 0 | 2
  Neutrophil count decreased | 0 | 2 | 1 | 3
  Platelet count decreased | 1 | 3 | 1 | 2
  White blood cell count decreased | 0 | 2 | 0 | 2
  Hypoalbuminaemia | 0 | 2 | 0 | 1
  Hypocalcaemia | 0 | 1 | 0 | 1
  Hypokalaemia | 0 | 3 | 0 | 2
  Hypomagnesaemia | 1 | 2 | 0 | 1
  Hyponatraemia | 0 | 2 | 0 | 2
  Hypophosphataemia | 0 | 1 | 0 | 0
  Proteinuria | 1 | 0 | 0 | 0
  Hyperthyroidism | 0 | 0 | 0 | 1
  Amylase increased | 0 | 0 | 1 | 1
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 1
  Lipase increased | 0 | 0 | 0 | 1

6. Primary Outcome: Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Dose Expansion Phase
Description: The OR is defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target lesions (TLs) and non-target lesions (NTLs), any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the sum of the diameters (SoD) of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. Percentage of participants with OR is reported.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: The intent-to treat (ITT) population included all participants who were randomized and received any study drugs and were analyzed according to randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Percentage of Participants | 29.0 [18.2 to 41.9] | 21.1 [9.6 to 37.3] | 32.9 [22.1 to 45.1]
Statistical Analysis 1: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel; Test type: Superiority; p = 0.3614, Cochran-Mantel-Haenszel — Nominal P-value for comparison of treatment groups obtained from Cochran-Mantel-Haenszel-test was stratified by cluster of differentiation 73 (CD73) level; Rate difference = -8.0, 95% CI 2-sided [-27.6 to 12.1]; 80% Confidence Interval 2-Sided: -20.9 to 5.2
Statistical Analysis 2: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel; Test type: Superiority; p = 0.6503, Cochran-Mantel-Haenszel — Nominal P-value for comparison of treatment groups obtained from Cochran-Mantel-Haenszel-test was stratified by CD73 level; Rate difference = 3.8, 95% CI 2-sided [-13.2 to 20.7]; 80% Confidence Interval 2-Sided: -7.4 to 15.0

7. Secondary Outcome: Number of Participants With TEAEs and TESAEs in Dose Expansion Phase
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 172.1 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants
  Any TEAEs | 62 | 37 | 70
  Any TESAEs | 34 | 24 | 37

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Dose Expansion Phase
Description: as for outcome 3
Time Frame: Day 1 through 172.1 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants
  Hypothermia | 0 | 0 | 1
  Pyrexia | 15 | 12 | 21
  Dyspnoea | 7 | 6 | 8
  Dyspnoea exertional | 1 | 1 | 2
  Hypertension | 2 | 3 | 11
  Hypotension | 3 | 4 | 4
  Orthostatic hypotension | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal ECG Parameters Reported as TEAEs in Dose Expansion Phase
Description: Number of participants with abnormal ECG parameters reported as TEAEs are reported.
Time Frame: Day 1 through 172.1 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants
  Supraventricular tachycardia | 0 | 1 | 0
  Tachycardia | 2 | 3 | 3

10. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Dose Expansion Phase
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Time Frame: Day 1 through 172.1 weeks (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants
  Anaemia | 17 | 14 | 28
  Febrile neutropenia | 0 | 1 | 3
  Leukocytosis | 1 | 0 | 1
  Leukopenia | 1 | 2 | 3
  Lymphopenia | 2 | 0 | 2
  Neutropenia | 22 | 15 | 16
  Thrombocytopenia | 6 | 7 | 13
  Thrombocytosis | 2 | 0 | 1
  Hyperthyroidism | 0 | 0 | 3
  Hypothyroidism | 0 | 0 | 7
  Hypertransaminasaemia | 0 | 1 | 0
  Alanine aminotransferase decreased | 1 | 0 | 0
  Alanine aminotransferase increased | 8 | 9 | 16
  Amylase increased | 1 | 0 | 1
  Aspartate aminotransferase increased | 11 | 8 | 15
  Blood albumin decreased | 1 | 0 | 0
  Blood alkaline phosphatase increased | 3 | 2 | 8
  Blood bilirubin increased | 3 | 3 | 2
  Blood creatinine increased | 2 | 0 | 8
  Blood glucose increased | 0 | 2 | 0
  Blood lactate dehydrogenase increased | 1 | 0 | 3
  Blood magnesium decreased | 0 | 1 | 0
  Blood oestrogen decreased | 0 | 1 | 0
  Gamma-glutamyltransferase increased | 6 | 1 | 8
  Haemoglobin decreased | 0 | 0 | 1
  International normalised ratio increased | 0 | 0 | 1
  Lipase increased | 0 | 1 | 2
  Liver function test increased | 1 | 0 | 0
  Lymphocyte count decreased | 4 | 2 | 6
  Neutrophil count | 0 | 0 | 1
  Neutrophil count decreased | 19 | 8 | 24
  Platelet count decreased | 13 | 9 | 20
  Troponin I increased | 1 | 0 | 0
  White blood cell count decreased | 6 | 6 | 10
  White blood cell count increased | 0 | 1 | 0
  Hyperglycaemia | 4 | 2 | 6
  Hyperkalaemia | 1 | 1 | 1
  Hypoalbuminaemia | 3 | 2 | 6
  Hypocalcaemia | 2 | 2 | 3
  Hypoglycaemia | 0 | 0 | 2
  Hypokalaemia | 4 | 2 | 8
  Hypomagnesaemia | 4 | 3 | 6
  Hyponatraemia | 8 | 0 | 3
  Hypophosphataemia | 1 | 0 | 0
  Hypovolaemia | 1 | 0 | 0
  Iron deficiency | 0 | 0 | 1
  Type 2 diabetes mellitus | 0 | 1 | 0
  Proteinuria | 0 | 1 | 1

11. Secondary Outcome: Percentage of Participants With OR According to RECIST v1.1 in Dose Escalation Phase
Description: The OR is defined as best overall response of confirmed CR or confirmed PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. Percentage of participants with OR is reported.
Time Frame: Baseline (Days -28 to -1) through 24.5 months (maximum observed duration)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Percentage of Participants | 0 [NA to NA] — There was zero responder in this cohort, so 95% confidence interval (CI) could not be calculated. | 14.3 [0.4 to 57.9] | 0 [NA to NA] — There was zero responder in this cohort, so 95% CI could not be calculated. | 12.5 [0.3 to 52.7]

12. Secondary Outcome: Percentage of Participants With Disease Control (DC) According to RECIST v1.1 in Dose Escalation Phase
Description: The DC is defined as confirmed CR, PR, or stable disease (SD) (maintained for >=8 weeks). The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis <10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from date of first documentation. The SD is defined as neither sufficient shrinkage of TLs to qualify for PR nor sufficient increase of TLs to qualify for progressive disease (PD), taking as reference the smallest SoD while on study, and no new lesions. The PD is defined as at least a 20% increase in SoD of TLs, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of SoD, or unequivocal progression of existing NTLs, or the appearance of new lesion/s. Percentage of participants with DC is reported.
Time Frame: Baseline (Days -28 to -1) through 24.5 months (maximum observed duration)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX
Number analyzed (Participants) | 7 | 7 | 3 | 8
Percentage of Participants | 42.9 [9.9 to 81.6] | 71.4 [29.0 to 96.3] | 66.7 [9.4 to 99.2] | 62.5 [24.5 to 91.5]

13. Secondary Outcome: Number of Participants With Overall Survival Events in Dose Expansion Phase
Description: The overall survival is defined as the time from the randomization until death due to any cause. For participants who were alive at the time of data cut off, overall survival was censored on the last date when participants were known to be alive. The overall survival is assessed using the Kaplan-Meier method. The number of participants with overall survival events (deaths) is reported.
Time Frame: Baseline (Days -28 to -1) through 38.7 months (maximum observed duration)
Population: The ITT population included all participants who were randomized and received any amount of study drugs and were analyzed according to randomized treatment assignment.
Measure: Number; unit: Participants with event
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants with event | 47 | 32 | 53
Statistical Analysis 1: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 1.260, 95% CI 2-sided [0.790 to 1.983] — Hazard ratio for comparison between treatment groups obtained from Cox Proportional Hazards model stratified by CD73 level with ties handled by the Efron method
Statistical Analysis 2: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.750, 95% CI 2-sided [0.498 to 1.131] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Overall Survival in Dose Expansion Phase
Description: The overall survival is defined as the time from the randomization until death due to any cause. For participants who were alive at the time of data cut off, overall survival was censored on the last date when participants were known to be alive. The overall survival is assessed using the Kaplan-Meier method.
Time Frame: Baseline (Days -28 to -1) through 38.7 months (maximum observed duration)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Months | 10.8 [8.2 to 13.2] | 8.9 [6.9 to 11.5] | 12.9 [10.1 to 15.3]

15. Secondary Outcome: Number of Participants With Progression-free Survival Events According to RECIST v1.1 in Dose Expansion Phase
Description: Progression-free survival (PFS) is defined as the time from randomization until the first documentation of a PD or death due to any cause, whichever occurred first, regardless of whether the participant received subsequent anticancer treatment prior to progression. The PD is defined as at least a 20% increase in sum of the diameters of target lesions, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of sum of the diameters, or unequivocal progression of existing non-target lesions, or the appearance of new lesion/s. Participants who had no documented progression and were still alive at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST v1.1 assessment. The PFS is assessed using the Kaplan-Meier method. The number of participants with PFS events is reported.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: as for outcome 13
Measure: Number; unit: Participants with event
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Participants with event | 43 | 32 | 51
Statistical Analysis 1: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 1.160, 95% CI 2-sided [0.726 to 1.837] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Dose-expansion, Gemcitabine + Nab-paclitaxel vs Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.719, 95% CI 2-sided [0.468 to 1.105] — [estimate comment as in outcome 13, analysis 1]

16. Secondary Outcome: Progression-free Survival According to RECIST v1.1 in Dose Expansion Phase
Description: The PFS is defined as the time from randomization until the first documentation of a PD or death due to any cause, whichever occurred first, regardless of whether the participant received subsequent anticancer treatment prior to progression. The PD is defined as at least a 20% increase in sum of the diameters of target lesions, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of sum of the diameters, or unequivocal progression of existing non-target lesions, or the appearance of new lesion/s. Participants who had no documented progression and were still alive at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST v1.1 assessment. The PFS is assessed using the Kaplan-Meier method.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Months | 6.7 [5.5 to 9.0] | 5.6 [3.5 to 7.5] | 7.5 [5.5 to 10.9]

17. Secondary Outcome: Duration of Response (DoR) According to RECIST v1.1 in Dose Expansion Phase
Description: The DoR is defined as the time from the first documentation of an OR until the first documentation of a PD or death due to any cause, whichever occurs first. The OR is defined as best overall response of confirmed CR or PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The PD is defined as at least a 20% increase in SoD of TLs, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of SoD, or unequivocal progression of existing NTLs, or the appearance of new lesion/s. The DoR is assessed using the Kaplan-Meier method.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: The ITT population included all participants who were randomized and received any amount of study drugs and were analyzed according to randomized treatment assignment. The DoR is assessed for only those participants who had OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 18 | 8 | 23
Months | 7.2 [4.9 to NA] — Upper limit of 95% CI was not calculated because an insufficient number of participants had event. | 12.9 [2.2 to NA] — Upper limit of 95% CI was not calculated because an insufficient number of participants had event. | 9.5 [5.7 to 12.0]

18. Secondary Outcome: Percentage of Participants With DC According to RECIST v1.1 in Dose Expansion Phase
Description: The DC is defined as confirmed CR, PR, or stable disease (SD) (maintained for >=8 weeks). The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis <10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from date of first documentation. The SD is defined as neither sufficient shrinkage of TLs to qualify for PR nor sufficient increase of TLs to qualify for PD, taking as reference the smallest SoD while on study, and no new lesions. The PD is defined as at least a 20% increase in SoD of TLs, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of SoD, or unequivocal progression of existing NTLs, or the appearance of new lesion/s. Percentage of participants with DC is reported.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 62 | 38 | 70
Percentage of Participants | 66.1 [53.0 to 77.7] | 73.7 [56.9 to 86.6] | 75.7 [64.0 to 85.2]

19. Secondary Outcome: Percentage of Participants With OR According to RECIST v1.1 by CD73 Expression at Baseline in Dose Expansion Phase
Description: The OR is defined as best overall response of confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis <10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The OR is assessed by cluster of differentiation 73 (CD73) expression level either low or high at baseline. The CD73 low is defined as no CD73 expression in tumor cells or <50% of tumor cells with 2+ or 3+ intensity and CD73 high is defined as CD73 expression with 2+ or 3+ intensity in >=50% of tumor cells.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: The ITT population included all participants who were randomized and received any amount of study drugs and were analyzed according to randomized treatment assignment. Here, "number of participants analyzed" (N) signified those participants who had high or low levels of CD73.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Gemcitabine + Nab-paclitaxel: CD73 Level = High: In dose-expansion phase, participants with 1L metastatic disease and high CD73 levels received IV infusions of chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High: In dose-expansion phase, participants with 1L metastatic disease and high CD73 levels received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High: In dose-expansion phase, participants with 1L metastatic disease and high CD73 levels received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Gemcitabine + Nab-paclitaxel: CD73 Level = Low: In dose-expansion phase, participants with 1L metastatic disease and low CD73 levels received IV infusions of chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low: In dose-expansion phase, participants with 1L metastatic disease and low CD73 levels received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low: In dose-expansion phase, participants with 1L metastatic disease and low CD73 levels received IV infusions of oleclumab 3000 mg every 2 weeks for 4 doses, then Q4W in combination with durvalumab 1500 mg Q4W plus chemotherapy of gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, both on Days 1, 8, and 15 and then repeated on Q4W schedule until disease progression, intolerable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
Arm/Group | Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low
Number analyzed (Participants) | 46 | 27 | 51 | 16 | 11 | 19
Percentage of Participants | 23.9 [12.6 to 38.8] | 22.2 [8.6 to 42.3] | 31.4 [19.1 to 45.9] | 43.8 [19.8 to 70.1] | 18.2 [2.3 to 51.8] | 36.8 [16.3 to 61.6]
Statistical Analysis 1: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Rate difference = -1.7, 95% CI 2-sided [-25.2 to 21.9]
Statistical Analysis 2: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Rate difference = 7.5, 95% CI 2-sided [-12.6 to 27.0]
Statistical Analysis 3: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Rate difference = -25.6, 95% CI 2-sided [-58.3 to 13.9]
Statistical Analysis 4: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Rate difference = -6.9, 95% CI 2-sided [-39.1 to 26.6]

20. Secondary Outcome: Number of Participants With Overall Survival Events by CD73 Expression at Baseline in Dose Expansion Phase
Description: The overall survival is defined as the time from the randomization until death due to any cause. For participants who were alive at the time of data cut off, overall survival was censored on the last date when participants were known to be alive. The overall survival is assessed by CD73 expression level either low or high at baseline using the Kaplan-Meier method. The CD73 low is defined as no CD73 expression in tumor cells or <50% of tumor cells with 2+ or 3+ intensity and CD73 high is defined as CD73 expression with 2+ or 3+ intensity in >=50% of tumor cells. The number of participants with overall survival events (deaths) is reported.
Time Frame: Baseline (Days -28 to -1) through 38.7 months (maximum observed duration)
Population: as for outcome 19
Measure: Number; unit: Participants with event
Arm/Group | Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low
Number analyzed (Participants) | 46 | 27 | 51 | 16 | 11 | 19
Participants with event | 37 | 22 | 39 | 10 | 10 | 14
Statistical Analysis 1: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Hazard Ratio (HR) = 1.173, 95% CI 2-sided [0.676 to 1.985] — Hazard ratio for comparison between treatment groups obtained from Cox Proportional Hazards model with ties handled by the Efron method
Statistical Analysis 2: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Hazard Ratio (HR) = 0.605, 95% CI 2-sided [0.377 to 0.968] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 3: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Hazard Ratio (HR) = 1.549, 95% CI 2-sided [0.622 to 3.917] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 4: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Hazard Ratio (HR) = 1.472, 95% CI 2-sided [0.638 to 3.576] — [estimate comment as in outcome 20, analysis 1]

21. Secondary Outcome: Overall Survival by CD73 Expression at Baseline in Dose Expansion Phase
Description: The overall survival is defined as the time from the randomization until death due to any cause. For participants who were alive at the time of data cut off, overall survival was censored on the last date when participants were known to be alive. The overall survival is assessed by CD73 expression level either low or high at baseline using the Kaplan-Meier method. The CD73 low is defined as no CD73 expression in tumor cells or <50% of tumor cells with 2+ or 3+ intensity and CD73 high is defined as CD73 expression with 2+ or 3+ intensity in >=50% of tumor cells.
Time Frame: Baseline (Days -28 to -1) through 38.7 months (maximum observed duration)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low
Number analyzed (Participants) | 46 | 27 | 51 | 16 | 11 | 19
Months | 9.9 [6.8 to 12.2] | 7.9 [4.2 to 9.7] | 12.1 [8.6 to 15.0] | 22.2 [10.2 to 33.6] | 16.0 [5.7 to 22.6] | 16.1 [10.3 to 21.0]

22. Secondary Outcome: Number of Participants With Progression-free Survival Events According to RECIST v1.1 by CD73 Expression at Baseline in Dose Expansion Phase
Description: PFS: Time from randomization until first documentation of PD/death due to any cause, whichever occurred first, regardless of whether participant received subsequent anticancer treatment prior to progression. PD:>=20% increase in SoD of TLs and an absolute increase of >= 5 mm of SoD/unequivocal progression of existing NTLs/appearance of new lesion. Participants who had no documented progression and were still alive at the time of analysis were censored at time of latest date of assessment from their last evaluable RECIST v1.1 assessment. PFS is assessed by CD73 expression level either low/high at baseline using Kaplan-Meier method. CD73 low: No CD73 expression in tumor cells/<50% of tumor cells with 2+/3+ intensity. CD73 high: CD73 expression with 2+/3+ intensity in >=50% of tumor cells. Number of participants with PFS events is reported.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: as for outcome 19
Measure: Number; unit: Participants with event
Arm/Group | Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low
Number analyzed (Participants) | 46 | 27 | 51 | 16 | 11 | 19
Participants with event | 35 | 23 | 39 | 8 | 9 | 12
Statistical Analysis 1: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Hazard Ratio (HR) = 1.004, 95% CI 2-sided [0.584 to 1.693] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = High vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High; Test type: Superiority; Hazard Ratio (HR) = 0.598, 95% CI 2-sided [0.366 to 0.973] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 3: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Hazard Ratio (HR) = 1.933, 95% CI 2-sided [0.716 to 5.437] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 4: Comparison: Gemcitabine + Nab-paclitaxel: CD73 Level = Low vs Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low; Test type: Superiority; Hazard Ratio (HR) = 1.374, 95% CI 2-sided [0.550 to 3.707] — [estimate comment as in outcome 20, analysis 1]

23. Secondary Outcome: Progression-free Survival According to RECIST v1.1 by CD73 Expression at Baseline in Dose Expansion Phase
Description: The PFS is defined as the time from randomization until the first documentation of a PD or death due to any cause, whichever occurred first, regardless of whether the participant receives subsequent anticancer treatment prior to progression. The PD is defined as at least a 20% increase in SoD of TLs, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of SoD, or unequivocal progression of existing NTLs, or the appearance of new lesion/s. Participants who had no documented progression and were still alive at time of analysis were censored at time of latest date of assessment from their last evaluable RECIST v1.1 assessment. PFS is assessed by CD73 expression level either low/high at baseline using Kaplan-Meier method. CD73 low: No CD73 expression in tumor cells/<50% of tumor cells with 2+/3+ intensity. CD73 high: CD73 expression with 2+/3+ intensity in >=50% of tumor cells.
Time Frame: Baseline (Days -28 to -1) through 36.1 months (maximum observed duration)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = High | Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel: CD73 Level = Low | Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel: CD73 Level = Low
Number analyzed (Participants) | 46 | 27 | 51 | 16 | 11 | 19
Months | 5.6 [3.7 to 7.4] | 5.2 [1.9 to 6.3] | 5.5 [4.4 to 9.3] | 10.5 [6.9 to NA] — Upper limit of 95% CI was not calculated because an insufficient number of participants had event. | 7.6 [3.3 to 11.2] | 10.9 [5.7 to 13.2]

24. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to Oleclumab
Description: Number of participants with positive ADA to oleclumab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with <16 weeks between first and last positive). Treatment-boosted ADA is defined as baseline ADA positive titer that was boosted to a 4-fold or higher level following drug administration.
Time Frame: Day 1 through 172.1 weeks (Pre-dose on Cycle [C] 1 Day [D] 1, C2D1, C3D1, Day 1 of every 3 cycles starting with C5, through 12 weeks post last dose of oleclumab)
Population: The ADA evaluable oleclumab population included all participants who received oleclumab, analyzed according to the treatment they actually received, and who had a non-missing baseline ADA result and at least one non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 6 | 7 | 3 | 7 | 31 | 63
Participants
  ADA positive at baseline | 0 | 0 | 0 | 0 | 0 | 0
  ADA positive post-baseline | 1 | 0 | 0 | 1 | 1 | 0
  Persistent Positive | 1 | 0 | 0 | 1 | 0 | 0
  Transient Positive | 0 | 0 | 0 | 0 | 1 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Positive ADA to Durvalumab
Description: Number of participants with positive ADA to durvalumab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with <16 weeks between first and last positive). Treatment-boosted ADA is defined as baseline ADA positive titer that was boosted to a 4-fold or higher level following drug administration.
Time Frame: Day 1 through 128 weeks (Pre-dose on C1D1, C2D1, C3D1, Day 1 of every 3 cycles starting with C5, through 12 weeks post last dose of durvalumab)
Population: The ADA evaluable durvalumab population included all participants who received durvalumab, analyzed according to the treatment they actually received, and who had a non-missing baseline ADA result and at least one non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 6 | 7 | 3 | 7 | 60
Participants
  ADA positive at baseline | 0 | 0 | 0 | 0 | 2
  ADA positive post-baseline | 1 | 0 | 0 | 2 | 0
  Persistent Positive | 1 | 0 | 0 | 2 | 0
  Transient Positive | 0 | 0 | 0 | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Serum Concentrations of Oleclumab
Description: Serum concentrations of oleclumab are reported.
Time Frame: Ten minutes (mins) (± 5 mins) post end of infusion (EOI), approximately 1 hour (+ 15 mins) after start of infusion on C1D1, C3D1, and C5D1; and pre-dose on C3D1 and C5D1
Population: Pharmacokinetic (PK) evaluable oleclumab population included all participants who received at least one dose of oleclumab and who had at least one reportable PK concentration. Here, number analyzed (n) denotes those participants who were analyzed for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 7 | 7 | 3 | 8 | 38 | 70
μg/mL
  C1D1 (EOI): number analyzed (Participants) | 7 | 7 | 3 | 7 | 37 | 70
  C1D1 (EOI) | 297.6 (25.70) | 710.2 (21.42) | 412.7 (11.12) | 734.6 (41.01) | 704.4 (30.28) | 725.9 (34.69)
  C3D1 (pre-dose): number analyzed (Participants) | 3 | 5 | 3 | 4 | 27 | 57
  C3D1 (pre-dose) | 128.6 (10.00) | 211.5 (73.40) | 134.3 (141.5) | 368.9 (2.461) | 164.8 (324.1) | 226.8 (70.41)
  C3D1 (EOI): number analyzed (Participants) | 2 | 5 | 3 | 4 | 25 | 57
  C3D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 870.3 (21.86) | 571.1 (15.75) | 1181 (24.97) | 893.0 (30.66) | 894.4 (39.22)
  C5D1 (pre-dose): number analyzed (Participants) | 1 | 3 | 0 | 4 | 20 | 45
  C5D1 (pre-dose) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 73.19 (130.2) |  | 235.7 (27.68) | 85.99 (192.0) | 116.4 (54.0)
  C5D1 (EOI): number analyzed (Participants) | 1 | 3 | 0 | 4 | 20 | 45
  C5D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 948.3 (44.90) |  | 1057 (14.88) | 852.8 (24.77) | 753.2 (41.32)

27. Secondary Outcome: Serum Concentrations of Durvalumab
Description: Serum concentrations of durvalumab are reported.
Time Frame: Ten mins (± 5 mins) post EOI, approximately 1 hour (+ 15 mins) after start of infusion on C1D1 and C5D1; and pre-dose on C2D1 and C5D1
Population: The PK evaluable durvalumab population included all participants who received at least one dose of durvalumab and who had at least one reportable PK concentration. Here, number of participants analyzed (N) indicates those participants who had adequate PK samples. Here, number analyzed (n) denotes those participants who were analyzed for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 7 | 7 | 3 | 8 | 70
μg/mL
  C1D1 (EOI) | 292.5 (11.72) | 374.5 (27.50) | 309.0 (11.58) | 380.7 (56.89) | 345.8 (324.2)
  C2D1 (pre-dose): number analyzed (Participants) | 5 | 6 | 3 | 7 | 61
  C2D1 (pre-dose) | 35.97 (51.44) | 14.39 (5129) | 50.52 (57.30) | 59.97 (176.7) | 86.20 (97.95)
  C5D1 (pre-dose): number analyzed (Participants) | 1 | 3 | 0 | 4 | 45
  C5D1 (pre-dose) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 74.52 (28.32) |  | 175.9 (43.50) | 137.9 (48.85)
  C5D1 (EOI): number analyzed (Participants) | 1 | 3 | 0 | 4 | 44
  C5D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 522.1 (46.72) |  | 664.5 (28.14) | 597.9 (23.40)

28. Secondary Outcome: Plasma Concentrations of Gemcitabine and Metabolite 2',2'-Difluorodeoxyuridine (dFdU)
Description: Plasma concentrations of gemcitabine and metabolite dFdU are reported.
Time Frame: Ten mins (± 5 mins) post EOI, approximately 30-40 mins after start of infusion on C1D1 and C4D1; and pre-dose on C4D1
Population: The PK evaluable gemcitabine population included all participants who received at least one dose of gemcitabine and who had at least one reportable PK concentration. Here, number analyzed (n) denotes those participants who were analyzed for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 7 | 7 | 57 | 38 | 70
ng/mL
  Gemcitabine C1D1 (EOI): number analyzed (Participants) | 7 | 7 | 54 | 36 | 65
  Gemcitabine C1D1 (EOI) | 3194 (64.74) | 4659 (67.41) | 3301 (192.0) | 3315 (135.4) | 4086 (148.9)
  Gemcitabine C4D1 (pre-dose): number analyzed (Participants) | 2 | 4 | 33 | 25 | 50
  Gemcitabine C4D1 (pre-dose) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point.
  Gemcitabine C4D1 (EOI): number analyzed (Participants) | 2 | 4 | 28 | 25 | 49
  Gemcitabine C4D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 3530 (48.11) | 1748 (236.5) | 1431 (446.3) | 2998 (151.3)
  dFdU C1D1 (EOI): number analyzed (Participants) | 7 | 7 | 54 | 36 | 65
  dFdU C1D1 (EOI) | 33700 (14.70) | 32160 (17.67) | 29510 (113.4) | 32350 (17.10) | 26300 (163.9)
  dFdU C4D1 (pre-dose): number analyzed (Participants) | 2 | 4 | 33 | 25 | 50
  dFdU C4D1 (pre-dose) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 434.6 (344.7) | 245.1 (361.5) | 149.9 (147.0) | 177.5 (170.0)
  dFdU C4D1 (EOI): number analyzed (Participants) | 2 | 4 | 28 | 25 | 49
  dFdU C4D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 34550 (35.37) | 23900 (189.1) | 21970 (130.3) | 27260 (43.07)

29. Secondary Outcome: Plasma Concentrations of Nab-paclitaxel
Description: Plasma concentrations of nab-paclitaxel are reported.
Time Frame: Ten mins (± 5 mins) post EOI, approximately 30-40 mins after start of infusion on C1D1 and C4D1; and pre-dose on C4D1
Population: The PK evaluable nab-paclitaxel population included all participants who received at least one dose of nab-paclitaxel and who had at least one reportable PK concentration. Here, number of participants analyzed (N) indicates those participants who had adequate PK samples. Here, number analyzed (n) denotes those participants who were analyzed for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
Number analyzed (Participants) | 7 | 7 | 60 | 38 | 70
ng/mL
  C1D1 (EOI): number analyzed (Participants) | 7 | 7 | 58 | 35 | 69
  C1D1 (EOI) | 1711 (80.37) | 2685 (63.55) | 2381 (105.2) | 2711 (81.67) | 2611 (142.0)
  C4D1 (pre-dose): number analyzed (Participants) | 2 | 4 | 35 | 24 | 47
  C4D1 (pre-dose) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point.
  C4D1 (EOI): number analyzed (Participants) | 2 | 4 | 31 | 24 | 48
  C4D1 (EOI) | NA (NA) — Per sponsor convention three observations > Lower Limit of Quantification were required as a minimum for a plasma concentration to be summarized. Otherwise, the statistics were not calculated at the time point. | 1474 (96.12) | 1825 (178.1) | 1445 (145.8) | 1747 (99.26)

ADVERSE EVENTS:
Time Frame: Day 1 through 172.1 weeks (maximum observed duration)
Arm/Group | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX | Dose-expansion, Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 7/7 | 7/7 | 3/3 | 8/8 | 47/62 | 32/38 | 53/70
Serious Adverse Events (participants affected / at risk) | 4/7 | 6/7 | 0/3 | 4/8 | 34/62 | 24/38 | 37/70
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 3/3 | 8/8 | 60/62 | 36/38 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=7) | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=7) | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX (N=3) | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX (N=8) | Dose-expansion, Gemcitabine + Nab-paclitaxel (N=62) | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel (N=38) | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=70)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 8 (9)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (4)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (6) | 1 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation, Oleclumab 1500 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=7) | Dose-escalation, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=7) | Dose-escalation, Oleclumab 1500 mg + Durvalumab + mFOLFOX (N=3) | Dose-escalation, Oleclumab 3000 mg + Durvalumab + mFOLFOX (N=8) | Dose-expansion, Gemcitabine + Nab-paclitaxel (N=62) | Dose-expansion, Oleclumab 3000 mg + Gemcitabine + Nab-paclitaxel (N=38) | Dose-expansion, Oleclumab 3000 mg + Durvalumab + Gemcitabine + Nab-paclitaxel (N=70)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (13) | 2 (3) | 1 (1) | 22 (37) | 14 (25) | 16 (36)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 8 (9) | 4 (9) | 7 (10)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (11) | 9 (10)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (6) | 7 (9) | 2 (2) | 6 (7) | 30 (33) | 25 (60) | 41 (54)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (10)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Oedema peripheral (General disorders) | 2 (4) | 3 (4) | 0 (0) | 2 (2) | 13 (15) | 12 (21) | 28 (41)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 1 (2) | 0 (0) | 1 (1) | 10 (14) | 10 (16) | 18 (26)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 2 (3) | 2 (3) | 1 (1) | 6 (8) | 7 (10) | 13 (24)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Portal vein occlusion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum purulent (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 3 (6)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 5 (7)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 1 (2) | 0 (0) | 17 (25) | 14 (15) | 27 (41)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 8 (9) | 9 (10) | 16 (22)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (6) | 0 (0) | 3 (3) | 11 (14) | 8 (9) | 15 (22)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 8 (9)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 8 (10)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood oestrogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (8) | 1 (1) | 8 (10)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 4 (11) | 2 (2) | 6 (8)
Neutrophil count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 3 (4) | 19 (41) | 8 (13) | 24 (49)
Platelet count decreased (Investigations) | 1 (2) | 3 (6) | 1 (2) | 2 (3) | 13 (39) | 9 (24) | 20 (50)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (4)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 7 (7) | 7 (8)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
White blood cell count decreased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 6 (19) | 6 (8) | 10 (19)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 16 (17) | 15 (58) | 21 (22)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 10 (12)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 6 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 6 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0) | 2 (3) | 4 (9) | 2 (3) | 8 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 4 (8) | 3 (3) | 6 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 8 (9) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 8 (10) | 7 (9) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (7) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 4 (4) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 8 (10) | 14 (19)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 10 (10)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 7 (7) | 6 (9)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 10 (10) | 5 (10) | 12 (13)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 3 (3) | 12 (13)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 11 (13) | 11 (12) | 13 (17)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 9 (11) | 11 (17) | 15 (17)
Polyneuropathy in malignant disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (9) | 7 (7)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 4 (5) | 11 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 6 (6) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 12 (12) | 11 (11) | 25 (26)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 6 (10) | 16 (18)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 6 (15) | 13 (14)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (17) | 12 (19)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cryoglobulinaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (3) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (7) | 10 (15)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orbital haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 12 (13) | 6 (7) | 13 (16)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 5 (5)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 10 (13) | 15 (21) | 18 (28)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (2) | 1 (1) | 5 (6) | 18 (26) | 14 (29) | 36 (63)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (8) | 2 (2) | 4 (5) | 26 (34) | 26 (70) | 41 (49)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 3 (5) | 7 (7)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 15 (21) | 12 (18) | 16 (23)

LIMITATIONS AND CAVEATS:
Dose escalation phase: Participants not enrolled in oleclumab 750 mg cohort. Dose expansion phase: Outcomes of mFOLFOX cohorts not included as enrollment was not opened. Non-compartmental PK data analysis were planned to be performed from each dose cohort if data allowed, but as sparse PK samples were collected, no non-compartmental PK parameters were calculated. Consequently, PK concentration time data only have been reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03611556/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03611556/SAP_001.pdf